CLINICAL TRIAL: NCT01342328
Title: Providing "Good Sleep" for ICU Sedation
Acronym: ASRV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Masimo Labs (Other)
Responsible Party: Principal Investigator, Mervyn Maze, MD, University of California, San Francisco
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 10-03906
Record Dates: First submitted 2010-12-07; First posted 2011-04-27 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Sleep Disorders
Keywords: Sleep disruption; Sleep hygiene; Sedative agents and sleep; Electroencephalography; REM sleep; Magnetoencephalography
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Hygiene | interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Placebo Comparator): For this arm, the volunteer subject will receive a saline infusion during the sleep session.
  Interventions: Other: Normal saline infusion
- Dexmedetomidine (DEX) (Experimental): For this arm, the volunteer subject will receive a DEX infusion for sedation during the sleep session.
  Interventions: Drug: Dexmedetomidine
- Propofol (Experimental): For this arm, the volunteer subject will receive a propofol infusion for sedation during the sleep session.
  Interventions: Drug: Propofol

INTERVENTIONS:
Other: Normal saline infusion — Normal saline infusion
  Arms: Control
Drug: Dexmedetomidine — Infusion of Dexmedetomidine will be administrated during the overnight sleep study. An initial target concentration of 0.25 ng/ml will be selected. After 5 min, the sedative point will be assessed and the concentration will be adjusted stepwise by increments and decrements of 0.05 ng/ml. This process will be repeated until the target sedative state is achieved. Using the Richmond Agitation Sedation Scale (RASS) infusion rates, using known pharmacokinetic parameters will be adjusted to achieve equivalent levels of sedation (RASS -3) for both DEX and propofol sessions.
  We aim to achieve an RASS of -3 so that the subjects are "moderately sedated". This state of sedation will be maintained for 3-4 hours.
  Other Names: Precedex; DEX
  Arms: Dexmedetomidine (DEX)
Drug: Propofol — For propofol, an initial concentration of 0.75 ng/ml will be targeted. Depending on the score achieved, the infusion rate will be increased or decreased every 5 min by 0.2 ng/ml until the target sedative state is achieved.
  Note that the target sedative state (RASS score of -3) is the same for both DEX and propofol sessions, with the investigator being unaware of which drug is being administered. To ensure the investigator is not aware of the type of drug being administered, all drug delivery systems will be covered.
  Intravenous drug delivery will be continued throughout the scanning period for 3-4 hours to maintain equivalent levels of sedation for both DEX and propofol.
  Other Names: Diprivan
  Arms: Propofol

SUMMARY:
Cognitive dysfunction, either alone or as an element in the syndrome of delirium, is a common occurrence with an incidence as high as 75% in intensive care unit (ICU) patients and can independently result in serious consequences including higher mortality rate. Delirium develops through a complex interaction between the patient's baseline vulnerability (risk factors) and precipitating factors such as disruption of sleep that may occur during hospitalization. While sedative-hypnotic agents that are used to facilitate hypnosis and the management of mechanically ventilated patients converge on the neural substrate that mediate endogenous sleep, they do so at different juncture points depending on its molecular mechanism of hypnotic action. Hypnotic agents that modulate the GABAA receptor converge at the level of the hypothalamus while α2 adrenergic agonists converge on sleep pathways within the brainstem. This translational project seeks to determine whether sedation mediated by activation of α2 adrenoceptors (dexmedetomidine) is more like natural sleep than that provided by a sedative agent that modulates the GABAA receptor (propofol). The investigators will examine volunteers who will be monitored continuously by electroencephalography (EEG) and whole-brain functional connectivity by magnetoencephalography (MEG) during each of three sleep stages, namely, that induced by dexmedetomidine, propofol, or saline (natural sleep, control). The two drug-induced sleep regimens will be compared to natural sleep using EEG and brain connectivity by MEG

DETAILED DESCRIPTION:
In this proposal the investigators seek to determine whether sedation mediated by activation of α2 adrenoceptors (dexmedetomidine) is more like natural sleep than that provided by a sedative agent that modulates the GABAA receptor (propofol), two common widely used sedative agents in ICU. Ten volunteers will be enrolled and each subject will be studied on three experimental sessions. Subjects will be randomized to receive a continuous infusion of either saline, dexmedetomidine (DEX), or propofol in each of the three sessions. By relying on clinical rating scales, the investigators ensure that the doses of DEX and propofol administered induce equisedative states before progressing to magnetoencephalography and electroencephalography data collection.

If the restorative and reparative benefits of sleep mitigate the development of cognitive dysfunction, this will result in shorter ICU length of stay for critically ill patients with a concomitant reduction in healthcare costs. Furthermore, it is possible that the restorative properties of sleep for the central nervous system can extend to the immune system with less infection and/or greater likelihood of survival from sepsis.

In this manner, our project will translate experimental data towards clinical practice and the adoption of rational and clinically supported interventions in the ICU that are likely to improve not only patient reported outcome measures, but also the chance of surviving critical illness.

Each experimental session will take a maximum of 7 hours (5 hours maximum for control sessions).

Sessions have to be separated by at least one week. Subjects will be enrolled for a minimum of 3 weeks (1 session on each week) and no more than 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer agreement and written informed consent
* Healthy female or male between 18 and 45 years of age
* Body Mass Index < 30 kg/m2
* Non-pregnant and non-lactating
* Normal airway anatomy (Mallampati class I)

Exclusion Criteria:

* Subject has a history of recent alcohol or drug abuse
* Subject is unable to communicate in English
* Subject is unwilling to meet fast guidelines (fast light meal or non-human milk for at least 8 hours, and clear liquids at least for 2 hours prior to induction of sedation on the day of the study)
* Subject has taken caffeine containing beverages less than 8 hours before study begins
* Subject is not able to avoid sleep for a minimum of 16 hours prior to testing
* Subject has a known allergy to either of the sedative-hypnotic drugs to be used in the study
* Subject has abnormal airway anatomy, including loose teeth
* Subject has any family history of complications from anesthesia
* Subject has history of sleep apnea
* Subject has any reported illness, upper respiratory tract infection, abnormal vital signs, or concerning findings on the physical exam for the past 6 weeks
* Subject has a positive urine pregnancy test
* Subject is unable to sleep supine.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2012-05; Primary Completion 2018-10-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Compare the electroencephalography features of sleep produced by three sleep-induced regimens | Data will be collected during patient's sleep, which will last 4hours.
  The investigators will evaluate the "power" in the delta rhythm range and amount of slow-wave-sleep
Compare the magnetoencephalography features of sleep produced by three sleep induced regimens | Data will be collected during patient's sleep, which will last 4hours.
  The investigators will evaluate the magnetoencephalography-defined brain connectivity

CONTACTS AND LOCATIONS:
Overall Officials: Mervyn Maze, MB, ChB, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States